CLINICAL TRIAL: NCT03353623
Title: A Randomized Controlled Single-Blind Crossover Trial on the Effects of Serious Games and Wearable Haptic Devices in the Rehabilitation of Children With Neuromotor Impairments
Brief Title: Immersive Virtual Environments and Wearable Haptic Devices in Rehabilitation of Children With Neuromotor Impairments
Acronym: SERIOUSGAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scuola Superiore Sant'Anna di Pisa (Other)
Collaborators: Unit of Developmental Neurorehabilitation, Pisa University Hospital (Unknown)
Responsible Party: Principal Investigator, Antonio Frisoli, Full Professor of Robotics and Mechanical Engineering, Scuola Superiore Sant'Anna di Pisa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: [SG]-CIV-IT-17-04-019324
Record Dates: First submitted 2017-11-15; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Cerebral Palsy; Dyspraxia
Keywords: Immersive Virtual Environments; Wearable Haptic Devices; Neuromotor Impairments; Rehabilitation; Serious Game; Randomized Controlled Trial
MeSH Terms: conditions — Cerebral Palsy; Apraxias

STUDY DESIGN:
Intervention Model Description: The investigators adopted a 2x2 crossover design (2-sequence, 2-period, 2-treatment crossover design, with sequences AB and BA): each participant received both conventional and VR-aided therapy for a period of 4 weeks per treatment (2 sessions per week of 45 minutes) assigned in a different order. A wash out period of 4 weeks was included before the second period of intervention started.
Who Masked: Outcomes Assessor
Masking Description: The study was masked only for the medical doctor who performed the motor assessments with clinical scales: she did not follow the rehabilitation sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ISG-Group (Immediate Serious Game) (Experimental): Children in the ISG-Group first participated in the VR-assisted rehabilitation, which consisted in 8 sessions with immersive virtual environment and wearable haptic devices, and were then crossed over and followed during an intended duration of 6 hours of conventional therapy.
  Interventions: Device: Serious Game; Other: Conventional Therapy
- DSG-Group (Delayed Serious Game) (Experimental): Children from DSG-Group were followed during an intended duration of 6 hours of conventional therapy before receiving VR-assisted rehabilitation with immersive virtual environment and wearable haptic devices.
  Interventions: Device: Serious Game; Other: Conventional Therapy

INTERVENTIONS:
Device: Serious Game — Serious Game (SG) refers to the use of immersive virtual environments and wearable haptic devices during the treatment. Two SG were specifically developed to allow a playful training of different, targeted Upper Limb (UL) movement based on typical rehabilitation exercises (reach-to-grasp, linear path tracking, hand orientation). The child interacts directly with a virtual environment through haptic feedback provided to his/her fingertips. In particular, "moneybox game" focused on pincer grasp and reaching tasks with pronation/supination od the hand while "marble labyrinth game" focused on pointing and tracking movements requiring both eye-hand and upper limb inter-joint coordination.
Other: Conventional Therapy — Conventional therapy (CONV) refers to the neurocognitive rehabilitation approach, with the purpose of improving pointing, tracking, reaching and grasping, and pronation/supination of the forearm. The therapeutic sessions were performed with the exception of the visual channel to ensure that the child focused his/her attention on tactile/kinesthetic information to complete the task. In particular, five different tasks have been proposed during the sessions: 1) recognize trajectories; 2) arm proprioception; 3) object manipulation; 4) recognize surfaces; 5) forearm orientation.

SUMMARY:
The investigators proposed a controlled, single-blind, unicentric, crossover, randomized, clinical trial to test the effects of immersive virtual environments and wearable haptic devices in the rehabilitation of children with neuromotor impairments. In addition, the proposed approach was compared with respect to conventional therapy.

A sample of 8 participants was randomly divided into 2 groups and they attended one of the two therapeutic approach for 4 weeks before crossing over and inverting the therapy. Between the two interventions, there was a wash out period of 4 weeks.

The investigators assessed motor abilities of the children with validated clinical scales and motion analysis before/after each phase of the study (T0: baseline, T1: after 4 weeks, T2: after 8 weeks, T3: after 16 weeks, and T4: up to 24 weeks).

DETAILED DESCRIPTION:
A Randomized Controlled Crossover Trial was designed to examine the usability and effectiveness of serious games and wearable haptic interfaces in rehabilitation of children with neuromotor impairments. The ethics board of Tuscany Region and the Italian Ministry of Health approved this study. All parents freely accepted the participation of their children in the study and provided written informed consent.

The investigators recruited eight patients, both male and female, 3 children with Cerebral Palsy (CP) and 5 children with Developmental Dyspraxia (DD) (mean age = 10,30±2,88 years), who were currently receiving conventional therapy at Unit of Developmental Neurorehabilitation, Maternal and Child Department, Pisa University Hospital, and eight Typically Developing children (TD, mean age = 9,60±2,61 years). All the patients were right-handed and they did not have previous experiences with Virtual Reality (VR) and/or haptic devices, while TD children have previously experienced with commercial video games.

Following recruitment, screening and consent and baseline assessments, participants are randomized to an order of VR-assisted rehabilitation (ISG-Group, Immediate Serious Games, or DSG-Group, Delayed Serious Games). Participants were setup in their first condition and were assessed at the end of the 4 week intervention. Participants were then set up in their second period for 4 weeks, again with assessment occurring at the end of the intervention. Among the two interventions, a wash out period of 4 weeks was inserted and children followed only cognitive therapy with no physical sessions.

The study protocol consisted of a total of 16 sessions with both VR-assisted and conventional rehabilitation (2 sessions per week for 4 weeks for 2 periods) and involved a familiarization and a training phase. The investigators adopted different established clinical scales for children with CP and DD in order to assess patients' abilities during the assessments. The investigators also selected metrics obtained from end-point (hand) kinematic data, including movement speed and accuracy, in order to have quantitative measurements of patients' motor abilities.

ELIGIBILITY:
Inclusion Criteria:

* a history of neuromotor disorders (CP or DD)
* a maximum age of 18 years
* a minimum ability to actively grasp an object
* the ability to understand simple instructions
* low to severe impairments of the upper limbs

Exclusion Criteria:

* epileptic patients
* severe deficit in sensory perception of upper limb
* severe visual impairments
* severe cognitive diseases

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Time Scores on Nine Hole Peg Test (9-HPT) for both Dominant and Non-Dominant Hands at 4, 8, 16 and 24 weeks | Baseline (T0), 4 weeks (T1), 8 weeks (T2), 16 weeks (T3), 24 weeks (T4)
  Nine Hole Peg Test (9-HPT) is a brief, standardized, quantitative test of upper extremity function. Both the dominant and non-dominant hands are tested twice. The child is seated at a table with a small, shallow container holding nine pegs and a wood or plastic block containing nine empty holes. On a start command when a stopwatch is started, the child picks up the nine pegs one at a time as quickly as possible, puts them in the nine holes, and, once they are in the holes, removes them again as quickly as possible one at a time, replacing them into the shallow container. The total time to complete the task is recorded.
Change From Baseline in Kinematic Metrics on Linear Path Tracking (LPT) and Reach-to-Grasp (RtG) Tasks for Dominant Hand at 4, 8, 16 and 24 weeks | Baseline (T0), 4 weeks (T1), 8 weeks (T2), 16 weeks (T3), 24 weeks (T4)
  The evaluation task consisted of two reach-to-grasp tasks requiring forearm pronation or supination and three linear path tracking (forward and sideways). For the RtG task, the child was asked to flip a card protruding from an horizontal support. For the LPT, the child was seated in front of a desk with the hand positioned, at rest, close to the body on the sagittal plane. Then a target was put on the desk (always at the same distance from the starting position) and the child was asked to reach the target by moving the hand along a straight path. All tasks were performed with the preferred arm at self selected speed. The investigators then extracted kinematic metrics (movement speed, accuracy and smoothness) from end-point (hand) kinematic data.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events according to the CTCAE v.4.0 | Up to 16 weeks
  The investigators referred to the following System Organ Class (SOC): Eye disorders, General disorders and administration site conditions, Nervous system disorders, Psychiatric disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Ilaria Bortone, PhD, Study Chair — PERCRO Laboratory, Scuola Superiore Sant'Anna, via L. Alamanno 13b, 56010 Ghezzano, Pisa, Italy
Locations (1):
- Unit of Developmental Neurorehabilitation, Maternal and Child Department, Pisa University Hospital, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Leonardis D, Solazzi M, Bortone I, Frisoli A. A 3-RSR Haptic Wearable Device for Rendering Fingertip Contact Forces. IEEE Trans Haptics. 2017 Jul-Sep;10(3):305-316. doi: 10.1109/TOH.2016.2640291. Epub 2016 Dec 15. PMID 28113306
- [Result] Bortone I, Leonardis D, Solazzi M, Procopio C, Crecchi A, Bonfiglio L, Frisoli A. Integration of serious games and wearable haptic interfaces for Neuro Rehabilitation of children with movement disorders: A feasibility study. IEEE Int Conf Rehabil Robot. 2017 Jul;2017:1094-1099. doi: 10.1109/ICORR.2017.8009395. PMID 28813967
- [Result] Leonardis, D., Solazzi, M., Bortone, I., & Frisoli, A. (2015, June). A wearable fingertip haptic device with 3 dof asymmetric 3-rsr kinematics. In World Haptics Conference (WHC), 2015 IEEE (pp. 388-393). IEEE.
- [Result] Bortone, I., Leonardis, D., Solazzi, M., Procopio, C., Crecchi, A., Briscese, L., ... & Frisoli, A. (2017). Serious Game and Wearable Haptic Devices for Neuro Motor Rehabilitation of Children with Cerebral Palsy. In Converging Clinical and Engineering Research on Neurorehabilitation II (pp. 443-447). Springer International Publishing.
- [Derived] Bortone I, Barsotti M, Leonardis D, Crecchi A, Tozzini A, Bonfiglio L, Frisoli A. Immersive Virtual Environments and Wearable Haptic Devices in rehabilitation of children with neuromotor impairments: a single-blind randomized controlled crossover pilot study. J Neuroeng Rehabil. 2020 Oct 28;17(1):144. doi: 10.1186/s12984-020-00771-6. PMID 33115487